CLINICAL TRIAL: NCT02776709
Title: Clinical Feasibility and Efficacy of a New Digital Single-operator Peroral Cholangiopancreatioscopy System: a Multicenter Registry
Brief Title: Feasibility of a Single-operator Peroral Cholangiopancreatioscopy System (SpyGlass)
Status: Withdrawn | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: University of Colorado, Denver (Other); University of California, Los Angeles (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); University of Utah (Other); Ochsner Health System (Other)
Responsible Party: Principal Investigator, Sri Komanduri, Director of Endoscopy, Northwestern University
Other Study IDs: STU00201104
Record Dates: First submitted 2016-05-12; First posted 2016-05-18 (Estimated); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Bile Duct Strictures; Common Bile Duct Stones
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Bile duct Stricture: Patients referred for the evaluation of indeterminate strictures.
  Interventions: Procedure: ERCP with cholangioscopy
- Common bile duct Stones: Patients referred for the removal of difficult stones.
  Interventions: Procedure: ERCP with cholangioscopy

INTERVENTIONS:
Procedure: ERCP with cholangioscopy

SUMMARY:
Cholangioscopy, or direct visualization of the bile ducts was first documented in the late 1970s and has made many advances over the last few decades. The advent of mother-baby scopes allowed for both diagnostic and therapeutic procedures, though the early scopes were often fragile, and cumbersome due to the need for two endoscopists. Ultraslim endoscopes later became popular as a method to digitally view the bile ducts, however, often needed guide-wire or balloon-assistance to allow for cannulation. Other disadvantages of these systems included limited steerability, and poor irrigation capabilities.

The advent of Spyglass, a single-operator peroral cholangioscopy method allowed for a fiberoptic, catheter-based system that could be easily used for diagnostic and therapeutic purposes in the biliary system. However, image quality was often lacking due to the fiberoptic technology. The new digital Spyglass system rectifies this inadequacy by introducing a digital sensor for better image quality, which will allow for better visualization and diagnosis of indeterminate strictures. Furthermore, modification of the scope platform allows for efficient use, reliable directionality of the scope tip, and improved ease of passage of accessories during therapeutic procedures such clearing stones or stent placement.

DETAILED DESCRIPTION:
All patients referred for the evaluation of indeterminate strictures or removal of difficult stones will be eligible for enrollment in the consortium. The PI or study coordinator will meet with the patient and discuss the study, its objectives, and obligations with each patient. After full disclosure, informed consent will be obtained.

Upon consent, basic demographics and data from prior procedures (when available) will be recorded. An endoscopist proficient in ERCP, with expertise in cholangioscopy, will perform the procedures using the Spyglass DS system with its associated components including biopsy forceps (SpyBiteTM) and other accessories as necessary. Procedure time, visual findings, number of biopsies taken, pathology, stone location, stone size, and method of stone clearance and adverse events will be recorded on data collection forms and transferred into a centralized password protected database. All patients will be followed for 6-12 months or surgery (stricture cohort) to assess accuracy or stone recurrence rates.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for the evaluation of indeterminate strictures or removal of difficult stones.

Exclusion Criteria:

* All patients who are unable or unwilling to give consent will not be included in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Formation of a multi-site prospective database of all patients referred for the evaluation of indeterminate strictures or removal of difficult stones.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Stone clearance rate | 6 months
  % of complete removal of bile duct stones

SECONDARY OUTCOMES:
Diagnostic accuracy for indeterminate bile duct strictures | 6 months
  Correlation of pathology with surgical specimen or 6month f/u

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - UCLA Medical Center, Los Angeles, California
  - University of Colorado, Denver, Denver, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Ochsner Medical Center, New Orleans, Louisiana
  - University of Utah, Salt Lake City, Utah